CLINICAL TRIAL: NCT01439334
Title: Multiple Behavior SBIRT Model of Drug Abuse in Primary Care
Brief Title: Multiple Behavior Screening, Brief Intervention and Referral to Treatment (SBIRT) Model of Drug Abuse in Primary Care
Acronym: SBIRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left UF
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2009-U-689; R01DA026028 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Drug Abuse
Keywords: Brief; Online; Image; Interactive; Young Adult; Primary Care
MeSH Terms: conditions — Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Online Program Brief (Experimental): Online Program Brief
  Interventions: Behavioral: MB-SBIRT (multiple behavior screening, brief intervention and referral to treatment) Online Program Brief
- Online Program Extended Length (Experimental): Online Program Extended Length
  Interventions: Behavioral: MB-SBIRT (multiple behavior screening, brief intervention and referral to treatment) Online Program Extended Length
- Control (Active Comparator): Control
  Interventions: Behavioral: MB-SBIRT (multiple behavior screening, brief intervention and referral to treatment) Control

INTERVENTIONS:
Behavioral: MB-SBIRT (multiple behavior screening, brief intervention and referral to treatment) Online Program Brief — Online prevention program using positive images
  Other Names: Online Program Brief
  Arms: Online Program Brief
Behavioral: MB-SBIRT (multiple behavior screening, brief intervention and referral to treatment) Online Program Extended Length — Online Program Extended Length
  Other Names: Online Program Extended Length
  Arms: Online Program Extended Length
Behavioral: MB-SBIRT (multiple behavior screening, brief intervention and referral to treatment) Control — Control
  Other Names: Control
  Arms: Control

SUMMARY:
The primary purpose of this research is to develop and evaluate the short-term efficacy of an innovative multiple behavior screening, brief intervention and referral to treatment (MB-SBIRT) model using social images and future self-images to simultaneously link and reduce prescription and other co-occurring drug use behaviors among emerging adults in a primary care setting serving a racially and economically diverse community. The long term objective of this research is to cost-effectively reduce prescription and illicit drug abuse, along with alcohol and tobacco consumption, and improve health-related quality of life among high-risk emerging adults often ignored in intervention research and services.

DETAILED DESCRIPTION:
Emerging adults are defined as young adults ages 18-25. These young people have the highest levels of prescription, illicit and licit drug consumption of any age group in the nation (Johnston, O'Malley, Bachman, & Schulenberg, 2007). While previous SBIRT models have typically targeted single health risks, such as problem alcohol or cigarette use, the proposed novel multiple behavior SBIRT model uses social and future images and a positive fitness theme to link co-morbid health risk behaviors and problems, and is therefore likely to be viewed by both patients and medical practitioners as appealing and feasible within standard primary care routines.

Objectives

1. Expanding and modifying existing social and future image screening and brief intervention content from our prior studies to include messages targeting prescription drug abuse and HIV/AIDS risk behaviors, as well as a referral to drug abuse assessment and treatment component;
2. Translating the modified and expanded multiple behavior SBIRT model content into two versions of the community-friendly computer-based program, i.e., one targeting one health promoting and four risk behaviors vs. another targeting four health promoting and four risk behaviors;
3. Conducting formative research on the modified content and format to ensure acceptability, quality, feasibility, accessibility, and potential effectiveness among target young adults and health care providers using expert panels, and target audience surveys; and
4. Conducting a three-group randomized trial pilot test with 3-month follow-up.

A three-group randomized trial pilot test will be conducted, with participating young adult patients randomized to receive either: 1) computer-based MB-SBIRT targeting one health promoting and four risk behaviors, 2) computer based MB-SBIRT targeting four health promoting and four risk behaviors, or 3) primary care as usual. This trial will determine the acceptability, quality, feasibility, and short-term (3-month) effects of the proposed computer delivered MB-SBIRT model.

ELIGIBILITY:
Inclusion Criteria:

* Understand English
* 18-25 Year old alcohol-drug using adults
* Attending the participating family care clinic

Exclusion Criteria:

* Can not understand English
* Not in age range
* Not attending participating clinic

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Change in prescription drug misuse, alcohol, cigarette and marijuana use consumption from baseline to 3 months follow up. | Baseline to 3 months follow up

SECONDARY OUTCOMES:
Change in frequency of health promoting behaviors from baseline to 3 months follow up. | Baseline to 3 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Chudley E Werch, PhD, Principal Investigator — Addictive & Health Behaviors Research Institute, University of Florida
Locations (1):
- Addictive & Health Behaviors Research Institute, University of Florida, Jacksonville, Florida, United States